CLINICAL TRIAL: NCT06272825
Title: Effectiveness of Virtual Reality in Patients With Symptomatic Knee Osteoarthritis
Brief Title: Virtual Reality in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-19/140
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Pain; Quality of Life
Keywords: Knee Osteoarthritis; virtual reaility; pain; Quality of Life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor will be different persons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to the conventional rehabilitation program at the hospital, virtual reality exercise will be applied in 15 sessions, 5 days a week.
  Interventions: Other: Virtual reality; Other: conventional rehabilitation
- Control group (Active Comparator): The conventional rehabilitation program at the hospital will be implemented in 15 sessions, 5 days a week.
  Interventions: Other: conventional rehabilitation

INTERVENTIONS:
Other: Virtual reality — VR-based exercise program will be applied in addition to the conventional rehabilitation program, 5 days a week for a total of 3 weeks.
  Arms: Experimental Group
Other: conventional rehabilitation — The conventional exercise program will include 20 minutes(Transcutaneous Electrical Nerve Stimulation) TENS with conventional method, 4 minutes continue ultrason, 20 minutes hot pack.

SUMMARY:
One of the main challenges facing the therapist in the treatment of adhesive capsulitis is to motivate the patient throughout conventional therapy. As noted in a recent review, individuals are more interested in leisure activities rather than performing repetitive tasks during therapy. Virtual reality (VR) is a three-dimensional computer-aided programme built with a system that creates virtual reality movements and generates a high amount of visual and sensory feedback during exercise. As a result, virtual reality (VR) has been used in many medical indications and has been shown to promote adherence to treatment by increasing patient motivation.

DETAILED DESCRIPTION:
Different VR systems have been shown to be effective in individuals with kinesiophobia as well as stroke patients. Virtual reality guided exercise is a proven method already used in stroke, Parkinson's, cerebral palsy rehabilitation, vestibular rehabilitation and orthopaedic rehabilitation. However, there is limited data on its effectiveness in patients with adhesive capsulitis. This randomized controlled study will contribute to the literature by investigating the effects of VR based exercises in individuals with AC

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic (>3 months) knee osteoarthritis between the ages of 40-85
* Kellgren and Lawrence Score ≥ 2 on knee radiograph
* Visual Analogue scale result VAS 4-8

Exclusion Criteria:

* Orthopedic surgery performed on the lower extremity
* Cognitive dysfunction (Mini Mental Test Score <23)
* Having received any treatment for knee osteoarthritis in the last 6 months
* Following any ongoing exercise program (tai chi, pilates, yoga, fitness)
* History of ligament and ligament injury around the knee

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-12-14 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels.
Visual Analog Scale | 3th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels.
Visual Analog Scale | 7th week
  Visual analog scale (VAS) was used for pain assessment. VAS is a 10-point Likert scale. Patients are asked to indicate their pain level, with 0 points being no pain, 5 points being moderate pain, and 10 points being unbearable pain. Increased scores indicate higher pain levels.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline
  WOMAC was used to assess disability in patients with knee osteoarthritis. The WOMAC assesses pain, stiffness and physical function and consists of 24 items. Total score is between 24 and 120 points. A low score indicates mild illness, a high score indicates severe illness.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3th week
  WOMAC was used to assess disability in patients with knee osteoarthritis. The WOMAC assesses pain, stiffness and physical function and consists of 24 items. Total score is between 24 and 120 points. A low score indicates mild illness, a high score indicates severe illness.
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 7th week
  WOMAC was used to assess disability in patients with knee osteoarthritis. The WOMAC assesses pain, stiffness and physical function and consists of 24 items. Total score is between 24 and 120 points. A low score indicates mild illness, a high score indicates severe illness.
Biodex Balance System | Baseline
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.
Biodex Balance System | 3th week
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.
Biodex Balance System | 7th week
  The balance assessment of the participants will be made with the Biodex Balance Systems device. During the measurement, patients will try to stay balanced on the device whose platform stability is adjusted.

SECONDARY OUTCOMES:
Short Form 36 (SF36) | Baseline
  In the study, quality of life will be evaluated using Short Form-36 (SF-36). SF-36 is not specific to any disease group. This scale consists of 36 questions; There are 8 subgroups: general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, and mental health. A high score is an indicator of good health.
Short Form 36 (SF36) | 3th week
  In the study, quality of life will be evaluated using Short Form-36 (SF-36). SF-36 is not specific to any disease group. This scale consists of 36 questions; There are 8 subgroups: general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, and mental health. A high score is an indicator of good health.
Short Form 36 (SF36) | 7th week
  In the study, quality of life will be evaluated using Short Form-36 (SF-36). SF-36 is not specific to any disease group. This scale consists of 36 questions; There are 8 subgroups: general health, physical function, physical role difficulty, pain, energy, social function, emotional role difficulty, and mental health. A high score is an indicator of good health.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asst Prof, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Kırşehir Ahi Evran University Faculty of Medicine, Kırşehir, City Center, Turkey (Türkiye)

REFERENCES:
- [Background] Wi, S. Y., & Kang, J. H. (2012). The effects of virtual reality interactive games on the balance ability of elderly women with knee osteoarthritis. Journal of Korean Society of Physical Medicine, 7(3), 387-393.
- [Background] Lin YT, Lee WC, Hsieh RL. Active video games for knee osteoarthritis improve mobility but not WOMAC score: A randomized controlled trial. Ann Phys Rehabil Med. 2020 Nov;63(6):458-465. doi: 10.1016/j.rehab.2019.11.008. Epub 2020 Jan 22. PMID 31981832
- [Background] Nambi G, Abdelbasset WK, Elsayed SH, Khalil MA, Alrawaili SM, Alsubaie SF. Comparative effects of virtual reality training and sensory motor training on bone morphogenic proteins and inflammatory biomarkers in post-traumatic osteoarthritis. Sci Rep. 2020 Sep 28;10(1):15864. doi: 10.1038/s41598-020-72587-2. PMID 32985509